CLINICAL TRIAL: NCT04696042
Title: Prospective Observational Study to Assess the Effectiveness and Safety of Lanreotide Autogel® in Patients With Locally Advanced or Metastatic Gastroenteropancreatic Neuroendocrine Tumors (GEP-NETs) in Asia Region
Brief Title: Asian Investigation of Lanreotide Autogel® in the Management of GEP-NETs
Acronym: AIM-NETs
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Samsung Medical Center (Other); Seoul St. Mary's Hospital (Other); Severance Hospital (Other); Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Changhoon Yoo, Assistant Professor, Asan Medical Center
Other Study IDs: AIM-NETs
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Neuroendocrine Tumors
Keywords: Neuroendocrine tumor; Somatostatin analogue
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lanreotide: Patients treated with lanreotide
  Interventions: Drug: Lanreotide autogel

INTERVENTIONS:
Drug: Lanreotide autogel — Lanreotide autogel 90-120 mcg, every 4 weeks

SUMMARY:
Lanreotide Autogel® has been established as a standard of care for patients with locally advanced or metastatic GEP-NETs based on the success of CLARINET trial. However, only few patients with Asian ethnicity were included in the trial.

According to the nationwide comprehensive study of patients with GEP-NET in Korea, hindgut primary NETs(Rectal) occured more frequently than western countries. However, small intestine or lung primary NET is relatively rare compared with western countries.1) Considering the clinical characteristics of GEP-NETs are distinct between the patients in Asian and Western countries, further evaluation on the efficacy and safety of Lanreotide Autogel® in Asian patients with GEP-NETs is needed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or female subject aged ≥18 years and legally capable to provide informed consent
* Functioning or non-functioning gastroenteropancreatic (GEP)-neuroendocrine tumor (NET) or unknown primary-NET
* Well differentiated tumor
* Grade (G) 1, G2 according to the 2017 World Health Organization (WHO) criteria
* Subject already treated with Lanreotide Autogel® for the period up to 5 months, according to local standard of care, prior to documentation into this study
* Use of Lanreotide autogel® monotherapy by local label (SmPC).
* Concomitant locoregional therapy such as surgery, RFA or TAE is allowed.

Exclusion Criteria:

* Parallel participation in an interventional study
* Lanreotide treatment for more than 5 months prior inclusion into the study
* Prior anti-proliferative medication with somatostatin analogue (e.g. Octreotide LAR).
* Concomitant anti-proliferative systemic medication/therapies for GEP-NET are not allowed.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: G1-2 GEP-NET patients who would be treated with lanreotide will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate at 2 years | 2 years
  Proportion of patients without tumor progression defined by RECIST version 1.1 at 2 years

SECONDARY OUTCOMES:
Progression-free survival | 2 years
  Time between lanreotide treatment initiation and disease progression or death
Response rates | 2 years
  Proportion of patients with tumor response by RECIST version 1.1
Disease control rates | 2 years
  Proportion of patients with tumor response and stable disease by RECIST version 1.1
Overall survival | 2 years
  Time between lanreotide treatment initiation and death due to any cause
Chromogranin A response | 2 years
  Change of serum chromogranin A levels during lanreotide treatment

CONTACTS AND LOCATIONS:
Overall Officials: Changhoon Yoo, Principal Investigator — Asan Medical Center
Locations (1):
- Changhoon Yoo, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gastrointestinal Pathology Study Group of Korean Society of Pathologists; Cho MY, Kim JM, Sohn JH, Kim MJ, Kim KM, Kim WH, Kim H, Kook MC, Park DY, Lee JH, Chang H, Jung ES, Kim HK, Jin SY, Choi JH, Gu MJ, Kim S, Kang MS, Cho CH, Park MI, Kang YK, Kim YW, Yoon SO, Bae HI, Joo M, Moon WS, Kang DY, Chang SJ. Current Trends of the Incidence and Pathological Diagnosis of Gastroenteropancreatic Neuroendocrine Tumors (GEP-NETs) in Korea 2000-2009: Multicenter Study. Cancer Res Treat. 2012 Sep;44(3):157-65. doi: 10.4143/crt.2012.44.3.157. Epub 2012 Sep 30. PMID 23091441
- [Background] Kim SJ, Kim JW, Oh DY, Han SW, Lee SH, Kim DW, Im SA, Kim TY, Heo DS, Bang YJ. Clinical course of neuroendocrine tumors with different origins (the pancreas, gastrointestinal tract, and lung). Am J Clin Oncol. 2012 Dec;35(6):549-56. doi: 10.1097/COC.0b013e31821dee0f. PMID 21659833
- [Background] Pavel M, O'Toole D, Costa F, Capdevila J, Gross D, Kianmanesh R, Krenning E, Knigge U, Salazar R, Pape UF, Oberg K; Vienna Consensus Conference participants. ENETS Consensus Guidelines Update for the Management of Distant Metastatic Disease of Intestinal, Pancreatic, Bronchial Neuroendocrine Neoplasms (NEN) and NEN of Unknown Primary Site. Neuroendocrinology. 2016;103(2):172-85. doi: 10.1159/000443167. Epub 2016 Jan 5. No abstract available. PMID 26731013
- [Background] Kang J, Yoo C, Hwang HS, Hong SM, Kim KP, Kim SY, Hong YS, Kim TW, Ryoo BY. Efficacy and safety of lanreotide in Korean patients with metastatic, well-differentiated gastroenteropancreatic-neuroendocrine tumors: a retrospective analysis. Invest New Drugs. 2019 Aug;37(4):763-770. doi: 10.1007/s10637-018-0710-x. Epub 2018 Dec 10. PMID 30536151
- [Background] Caplin ME, Pavel M, Cwikla JB, Phan AT, Raderer M, Sedlackova E, Cadiot G, Wolin EM, Capdevila J, Wall L, Rindi G, Langley A, Martinez S, Blumberg J, Ruszniewski P; CLARINET Investigators. Lanreotide in metastatic enteropancreatic neuroendocrine tumors. N Engl J Med. 2014 Jul 17;371(3):224-33. doi: 10.1056/NEJMoa1316158. PMID 25014687